CLINICAL TRIAL: NCT05978297
Title: Virtual Specialty Clinic for Fibromyalgia Care
Status: Active, not recruiting | Type: Observational
Sponsor: Swing Therapeutics, Inc. (Other)
Collaborators: Swing Care Provider Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: SC-001
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an ongoing, prospective, and retrospective cohort study of fibromyalgia patients who receive clinical care at Swing Care (a fibromyalgia virtual specialty clinic).

Deidentified data on demographics, clinical outcomes, patients' treatment engagement and preference, as well as patients' satisfaction are obtained and analyzed via retrospective and prospective chart review.

A waiver of informed consent has been approved by the reviewing Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of Swing Care between 1 Oct, 2022 and 1 Oct, 2027, who received clinical evaluations and/or treatments according to Swing Care's standard clinical care protocol.

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult fibromyalgia patients who receive clinical care at Swing Care.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Demographic and clinical data obtained via chart review [ Time Frame: 5 years ] | 01 Oct 2022 - 01 Oct 2027
  This is a clinic based registry of fibromyalgia patient outcomes from patients at the Swing Care clinic to be collected over time.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Chadwick, Principal Investigator — Swing Care
Locations (1):
- Swing Care, Covina, California, United States